CLINICAL TRIAL: NCT05861635
Title: Union Hospital Affiliated to Huazhong University of Science and Technology
Brief Title: The Study of Vidicizumab Combined With Tirelizumab in the Treatment of Breast Cancer With Low HER2 Expression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT22575
Record Dates: First submitted 2023-02-18; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disitamab Vedotin combined with Tislelizumab (Experimental): Subjects who meet the requirements of the protocol will receive neoadjuvant treatment, and the specific administration arrangement is as follows:
  Disitamab Vedotin, 2 mg/Kg, q2W, 8cycle Tislelizumab, 200mg, iv, q3W, 6cycle
  Interventions: Drug: Disitamab Vedotin combined with Tislelizumab

INTERVENTIONS:
Drug: Disitamab Vedotin combined with Tislelizumab — Subjects who meet the requirements of the protocol will receive neoadjuvant treatment, and the specific administration arrangement is as follows:
  Disitamab Vedotin, 2 mg/Kg, q2W, 8cycle Tislelizumab, 200mg, iv, q3W, 6cycle

SUMMARY:
To evaluate the efficacy and safety of vidicizumab combined with tirelizumab in the treatment of early high-risk or locally advanced breast cancer with low HER2 expression

DETAILED DESCRIPTION:
Studies have shown that vidicizumab has good efficacy and safety in advanced HER-2 low expression breast cancer. Vidicizumab combined with immunotherapy may be a new adjuvant treatment option for HER-2 low expression breast cancer patients. Therefore, we plan to carry out a clinical study to evaluate the efficacy, safety and tolerance of vidicizumab combined with tirelizumab during neoadjuvant therapy, in order to provide new treatment options for patients with breast cancer with HER-2 low expression in neoadjuvant therapy, improve their prognosis and improve their quality of life

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old, male or female;
2. Early or locally advanced breast cancer confirmed by pathology;
3. Lymph node positive or lymph node negative, ER and PR negative, T ≥ 2 or lymph node negative, ER positive or PR positive, T ≥ 5;
4. ECOG PS: 0-1; 5）Patients with low expression of HER-2: HER-2 IHC 1+or HER2 IHC 2+and ISH negative;

Exclusion Criteria:

1. Stage IV breast cancer;
2. Have received anti-tumor treatment or radiotherapy for any malignant tumor in the past five years, excluding cured cervical carcinoma in situ, skin basal cell carcinoma or squamous cell carcinoma;
3. At the same time, other clinical trials have received anti-tumor therapy. If the researcher judges that the patient cannot benefit from the researcher, other anti-tumor therapy can be ended.
4. The patient has undergone major surgery unrelated to breast cancer within 4 weeks before enrollment, or has not fully recovered from such surgery;
5. Previously received ADC drugs, immunosuppressants, anti-HER2 and other treatments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete remission (pCR) rate | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing Yao, Study Director — Xiehe Hospital
Locations (1):
- WuhanHU, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No